CLINICAL TRIAL: NCT01260311
Title: Post Marketing Surveillance To Assess The Safety And Efficacy Of Fesoterodine (Toviaz) On Filipino Patients Diagnosed With Over-Active Bladder
Brief Title: Post Marketing Surveillance Of Fesoterodine In Filipino Patients With Over Active Bladder
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A0221085
Record Dates: First submitted 2010-11-22; First posted 2010-12-15 (Estimated); Results first posted 2014-09-11 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Over Active Bladder
Keywords: Observational
MeSH Terms: interventions — fesoterodine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients prescribed with Fesoterodine: Patients diagnosed with Over-active bladder and prescribed with fesoterodine.
  Interventions: Drug: Fesoterodine

INTERVENTIONS:
Drug: Fesoterodine — Any dose of Fesoterodine
  Other Names: Toviaz

SUMMARY:
This is an observational study and will determine the safety profile of fesoterodine in Filipino patients prescribed the drug. This is in compliance with the requirements of the Philippine Food and Drug Administration.

DETAILED DESCRIPTION:
Sampling method is not applicable in this study. Only patients prescribed Fesoterodine will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Over-active bladder
* Prescribed with Fesoterodine

Exclusion Criteria:

* Hypersensitivity
* Urinary retention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Over-active bladder
Sampling Method: Non-Probability Sample
Enrollment: 508 (Actual)
Dates: Start 2011-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (37):
- Philippines (37):
  - Mary Johnston Hospital, Inc., Tondo, Manila
  - East Avenue Medical Center, Diliman, Quezon City, National Capital Region
  - The Medical City, Pasig, National Capital Region
  - St. Luke's Medical Center, Quezon City, National Capital Region
  - Private Clinic, Baguio City
  - Private Clinic, Batangas
  - Cebu Doctors Hospital, Osmena Blvd.,, Cebu
  - Private Clinic, City of Muntinlupa
  - Davao Doctors Hospital, Davao City
  - Davao Doctors Tower, Davao City
  - Davao Medical School Foundation Hospital, Davao City
  - Private Clinic, Davao City
  - Room 120, Davao Medical School Foundation Hospital, Davao City
  - Private Clinic, Ilocos Norte
  - Private Clinic, La Union
  - Private Clinic, Laguna
  - Lucena United Doctors Hospital, Lucena City
  - Makati Medical Center, Makati City
  - Private Clinic, Makati City
  - Room 314 Main Building, Makati City
  - VRPMC, Mandaluyong
  - Medical Center Manila, Manila
  - University of Sto. Tomas Hospital, Manila
  - Ospital ng Maynila Medical Center, Manila
  - Private Clinic, Manila
  - Santo Tomas University Hospital, Manila
  - Private Clinic, Nueva Ecija
  - Healthway Medical, The Block, Philippines
  - East Avenue Medical Center, Quezon
  - Private Clinic, Quezon
  - St. Luke's Medical Center, North Tower, CHBC, Quezon City
  - Private Clinic, Quezon City
  - Private Clinic, South Luzon
  - Central Luzon Doctor's Hospital, Tarlac City
  - Fatima Medical Center, Inc., Valenzuela
  - F.E.U. - Nicanor Reyes Medical Foundation Medical Center, West Fairview, Quezon City
  - Urology Clinic, Zamboanga City

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221085&StudyName=Post%20Marketing%20Surveillance%20Of%20Fesoterodine%20In%20Filipino%20Patients%20With%20Over%20Active%20Bladder

RESULTS

PARTICIPANT FLOW:
Groups:
- Fesoterodine Fumarate: Participants received fesoterodine fumarate (Toviaz) 4 milligram (mg) or 8 mg orally once daily, with use and dosage adjusted according to medical and therapeutic necessity.
Period: Overall Study
Arm/Group | Fesoterodine Fumarate
Started | 508
Completed | 381
Not Completed | 127
Not completed — Adverse Event | 11
Not completed — Lack of Efficacy | 4
Not completed — Lost to Follow-up | 25
Not completed — Withdrawal by Subject | 6
Not completed — Financial Constraints | 77
Not completed — Gone to Province | 2
Not completed — Medication Stopped | 1
Not completed — Fesoterodine Started Before Enrollment | 1

BASELINE CHARACTERISTICS:
Groups:
- Fesoterodine Fumarate: Participants received fesoterodine fumarate (Toviaz) 4 mg or 8 mg orally once daily, with use and dosage adjusted according to medical and therapeutic necessity.
Arm/Group | Fesoterodine Fumarate
Number analyzed (Participants) | 508
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 199
  Male | 309
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 64.1 (11.4)
Body Mass Index [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 24.1 (4.1)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 163.2 (10.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) by Seriousness, Severity and Relationship to Treatment
Description: Counts of participants who had treatment-emergent AEs (TEAEs), defined as newly occurring or worsening after first dose. Relatedness to fesoterodine fumarate (Toviaz) was assessed by the investigator. Participants with multiple occurrences of an AE within a category were counted once within the category. Seriousness of an AE was assessed under the criteria of serious adverse event (SAE). AE was assessed according to severity; mild (not causing any significant problem, dose adjustment not required), moderate (caused problem that does not interfere significantly with usual activities or the clinical status, dose adjustment needed due to AE) and severe (caused problem that interferes significantly with usual activities or the clinical status, study drug stopped due to AE).
Time Frame: Baseline up to 28 days after last dose
Population: Safety population defined as all participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Fesoterodine Fumarate
Number analyzed (Participants) | 508
participants
  Participants with AEs, all-causality | 21
  Participants with AEs, treatment-related | 19
  Participants with serious AEs, all-causality | 0
  Participants with serious AEs, treatment-related | 0
  Participants with severe AEs, all-causality | 2
  Participants with severe AEs, treatment-related | 2

2. Other Pre Specified Outcome: Number of Micturitions Per 24 Hours at Week 4 and Week 8
Description: Micturitions include episodes of voluntary micturition and episodes of Urgency Urinary Incontinence (UUI). UUI episodes were defined as those micturitions with Urinary Sensation Scale (USS) rating of 5 in the diary in participants with UUI at baseline. USS rating 5: Unable to hold; leak urine.
Time Frame: Week 4 and Week 8
Population: This efficacy outcome measure was removed in Protocol Amendment 1 and thus data was not collected.
Arm/Group | Fesoterodine Fumarate
Number analyzed (Participants) | 0

3. Other Pre Specified Outcome: Number of Urgency Episodes Per 24 Hours at Week 4 and Week 8
Description: Urgency episodes were defined as micturitions with USS rating of greater than or equal to (>=) 3. USS total range 1 to 5: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine.
Time Frame: Week 4 and Week 8
Population: This efficacy outcome measure was removed in Protocol Amendment 1 and thus data was not collected.
Arm/Group | Fesoterodine Fumarate
Number analyzed (Participants) | 0

4. Other Pre Specified Outcome: Number of UUI Episodes Per 24 Hours at Week 4 and Week 8
Description: UUI episodes were defined as those with USS rating of 5 in the diary. USS total range 1 to 5: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine.
Time Frame: Week 4 and Week 8
Population: This efficacy outcome measure was removed in Protocol Amendment 1 and thus data was not collected.
Arm/Group | Fesoterodine Fumarate
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Patient Perception of Bladder Condition (PPBC) at Week 4 and Week 8
Description: PPBC: a self-administered, single-item, questionnaire that asks participants to describe their perception of their bladder-related problems. The PPBC assessment is rated on a 6-point scale: 1=no problems at all, 2=some very minor problems, 3=some minor problems, 4=moderate problems, 5=severe problems, 6=many severe problems. Improvement is defined as negative change from baseline.
Time Frame: Week 4 and Week 8
Population: This efficacy outcome measure was removed in Protocol Amendment 1 and thus data was not collected.
Arm/Group | Fesoterodine Fumarate
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Fesoterodine Fumarate
Serious Adverse Events (participants affected / at risk) | 0/508
Other Adverse Events (participants affected / at risk) | 21/508
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fesoterodine Fumarate (N=508)
Palpitations (Cardiac disorders) | 1
Dry eye (Eye disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 10
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 1
Urinary tract infection (Infections and infestations) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Urinary retention (Renal and urinary disorders) | 2

LIMITATIONS AND CAVEATS:
The implementation of Protocol Amendment 1 led to removal of all primary efficacy outcome measures, therefore the efficacy outcome measures were not investigated or reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.